CLINICAL TRIAL: NCT02562859
Title: An Open-label Study to Compare the Oral Bioavailability of an Oral Tablet of GLPG1837 Relative to an Oral Suspension After Single-dose Intake in Healthy Subjects and to Evaluate the Effect of Food on the Oral Tablet
Brief Title: Oral Bioavailability of Solid Formulation of GLPG1837 With and Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GLPG1837-CL-103; 2015-002518-55 (EudraCT Number)
Record Dates: First submitted 2015-09-23; First posted 2015-09-29 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
MeSH Terms: interventions — GLPG1837; Suspensions; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GLPG1837 as oral suspension fasted (Experimental): Single dose of 500 mg GLPG1837 as oral suspension after an overnight fast
  Interventions: Drug: 500 mg GLPG1837 as oral suspension
- GLPG1837 as oral tablet fasted (Experimental): Single dose of 500 mg GLPG1837 as oral tablet after an overnight fast
  Interventions: Drug: 500 mg GLPG1837 as oral tablet
- GLPG1837 as oral tablet fed (Experimental): Single dose of 500 mg GLPG1837 as oral tablet after a high-fat high-calorie breakfast
  Interventions: Drug: 500 mg GLPG1837 as oral tablet

INTERVENTIONS:
Drug: 500 mg GLPG1837 as oral suspension — A single dose of 500 mg GLPG1837 administered as oral suspension
  Arms: GLPG1837 as oral suspension fasted
Drug: 500 mg GLPG1837 as oral tablet — A single dose of 500 mg GLPG1837 administered as oral tablet
  Arms: GLPG1837 as oral tablet fasted; GLPG1837 as oral tablet fed

SUMMARY:
The purpose of the study is to evaluate the amount of GLPG1837 and metabolite present in the blood (relative bioavailability) after a single oral administration of 500 mg GLPG1837 given as an oral suspension under fasted conditions as well as a tablet formulation under fasted and fed conditions, in male healthy subjects.

Also, the safety and tolerability of a single oral dose of 500 mg GLPG1837 given as an oral suspension under fasted conditions as well as a tablet formulation under fasted and fed conditions, will be assessed.

Twelve subjects will receive GLPG1837 on 3 occasions as single dose administrations: as an oral suspension fasted, as an oral tablet, fed and fasted. Treatment administrations will be separated by a wash-out period of at least 6 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, age 18-50 years
* BMI between 18-30 kg/m2

Exclusion Criteria:

* Any condition that might interfere with the procedures or tests in this study
* Drug or alcohol abuse
* Smoking

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The maximum observed concentration (Cmax) of GLPG1837 (metabolite) in plasma | Between Day 1 (predose) in period 1 (first dose of GLPG1837) and Day 4 (72h post dose) in period 3 (last dose of GLPG1837)
  To characterize and compare the maximum observed concentration (Cmax) of GLPG1837 (metabolite) in plasma in male healthy subjects after a single administration of an oral suspension versus an oral tablet formulation in fasted condition, and an oral tablet formulation in fasted versus fed condition
The concentration observed at 24 hours post dose (C24h) of GLPG1837 (metabolite) in plasma | Between Day 1 (predose) in period 1 (first dose of GLPG1837) and Day 2 (24h post dose) in period 3 (last dose of GLPG1837)
  To characterize and compare the concentration observed at 24 hours post dose (C24h) of GLPG1837 (metabolite) in plasma in male healthy subjects after a single administration of an oral suspension versus an oral tablet formulation in fasted condition, and an oral tablet formulation in fasted versus fed condition
The time of occurrence of Cmax (tmax) of GLPG1837 (metabolite) in plasma | Between Day 1 (predose) in period 1 (first dose of GLPG1837) and Day 4 (72h post dose) in period 3 (last dose of GLPG1837)
  To characterize and compare the time of occurrence of Cmax (tmax) of GLPG1837 (metabolite) in plasma in male healthy subjects after a single administration of an oral suspension versus an oral tablet formulation in fasted condition, and an oral tablet formulation in fasted versus fed condition
The area under the plasma concentration versus time curve (AUC) of GLPG1837 (metabolite) in plasma | Between Day 1 (predose) in period 1 (first dose of GLPG1837) and Day 4 (72h post dose) in period 3 (last dose of GLPG1837)
  To characterize and compare the area under the plasma concentration versus time curve of GLPG1837 (metabolite) in plasma in male healthy subjects after a single administration of an oral suspension versus an oral tablet formulation in fasted condition, and an oral tablet formulation in fasted versus fed condition
The apparent terminal half-life (t1/2) of GLPG1837 (metabolite) in plasma | Between Day 1 (predose) in period 1 (first dose of GLPG1837) and Day 4 (72h post dose) in period 3 (last dose of GLPG1837)
  To characterize and compare the apparent terminal half-life of GLPG1837 (metabolite) in plasma in male healthy subjects after a single administration of an oral suspension versus an oral tablet formulation in fasted condition, and an oral tablet formulation in fasted versus fed condition
The metabolite over GLPG1837 ratios in plasma | Between Day 1 (predose) in period 1 (first dose of GLPG1837) and Day 4 (72h post dose) in period 3 (last dose of GLPG1837)
  To characterize and compare the metabolite over GLPG1837 ratios in plasma in male healthy subjects after a single administration of an oral suspension versus an oral tablet formulation in fasted condition, and an oral tablet formulation in fasted versus fed condition

SECONDARY OUTCOMES:
Number of adverse events | Between Screening and 7 to 10 days after the last dose of GLPG1837
  To evaluate the safety and tolerability of a single dose of GLPG1837 administered as oral suspension fasted, oral tablet fasted versus fed in male healthy subjects in terms of number of adverse events (AEs) reported
Changes in vital signs as measured by heart rate, blood pressure and oral body temperature | Between Screening and 7 to 10 days after the last dose of GLPG1837
  To evaluate the safety and tolerability of a single dose of GLPG1837 administered as oral suspension fasted, oral tablet fasted versus fed in male healthy subjects in terms of changes in vital signs as measured by heart rate, blood pressure and oral body temperature reported
Changes in 12-lead ECG measures | Between Screening and 7 to 10 days after the last dose of GLPG1837
  To evaluate the safety and tolerability of a single dose of GLPG1837 administered as oral suspension fasted, oral tablet fasted versus fed in male healthy subjects in terms of changes in 12-ECG measures reported
Changes in physical exam measures | Between Screening and 7 to 10 days after the last dose of GLPG1837
  To evaluate the safety and tolerability of a single dose of GLPG1837 administered as oral suspension fasted, oral tablet fasted versus fed in male healthy subjects in terms of changes in physical examination reported
Changes in blood safety lab parameters | Between Screening and 7 to 10 days after the last dose of GLPG1837
  To evaluate the safety and tolerability of a single dose of GLPG1837 administered as oral suspension fasted, oral tablet fasted versus fed in male healthy subjects in terms of changes in blood safety lab parameters reported
Changes in urine safety lab parameters | Between Screening and 7 to 10 days after the last dose of GLPG1837
  To evaluate the safety and tolerability of a single dose of GLPG1837 administered as oral suspension fasted, oral tablet fasted versus fed in male healthy subjects in terms of changes in urine safety lab parameters reported

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV
Locations (1):
- SGS LSS Clinical Pharmacology Unit Antwerp, Antwerp, Antwerp, Belgium